CLINICAL TRIAL: NCT01559896
Title: The Effect of Egg Protein Hydrolysate on Arterial Stiffness in Overweight or Moderately Obese Subjects With Impaired Glucose Tolerance or Diabetes Type 2
Brief Title: Egg Protein Hydrolysate and Vascular Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NL36690.068.11
Record Dates: First submitted 2012-03-19; First posted 2012-03-21 (Estimated); Last update posted 2014-08-05 (Estimated); Status verified 2014-08

CONDITIONS: Arterial Stiffness; Dietary Modification; Impaired Glucose Tolerance; Type 2 Diabetes Mellitus
Keywords: egg protein hydrolysate
MeSH Terms: conditions — Glucose Intolerance; Diabetes Mellitus, Type 2 | interventions — Protein Hydrolysates

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- intervention and placebo (Experimental): Once in the study, 20 subjects will be randomly assigned to a group taking capsules containing 5 gr egg protein hydrolysate per day, and 20 to a group taking placebo capsules. The subjects consume the capsules during three consecutive days (period 1). Following a wash-out period of minimally four weeks, the treatments are crossed-over.
  Interventions: Dietary Supplement: protein hydrolysate capsules and placebo capsules

INTERVENTIONS:
Dietary Supplement: protein hydrolysate capsules and placebo capsules — Once in the study, 20 subjects will be randomly assigned to a group taking capsules containing 5 gr egg protein hydrolysate per day, and 20 to a group taking placebo capsules. The subjects consume the capsules during three consecutive days (period 1). Following a wash-out period of minimally four weeks, the treatments are crossed-over.

SUMMARY:
The incidence of type 2 diabetes mellitus (T2DM) is rapidly growing. Patients with T2DM are at increased risk of developing long term micro- and macrovascular complications. Subjects with impaired glucose tolerance (IGT) show increased blood glucose levels after an oral glucose load. These subjects have a markedly increased risk of later T2DM development.

T2DM development can be prevented or delayed by lifestyle modifications. To support lifestyle changes and reduce the risk of T2DM development, foods containing functional ingredients are being developed. An interesting functional ingredient is protein hydrolysate. An egg protein hydrolysate has been experimentally shown to improve endothelial function, to inhibit plasma angiotensin converting enzyme (ACE) and to reduce blood pressure in rats. Egg protein hydrolysate could thus be a interesting ingredient to treat the cardiovascular dysfunction associated with T2DM. In the present study, the effects of egg protein hydrolysate will be evaluated in subjects with overweight or moderate obesity and IGT or T2DM.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 70 years;
* male and female;
* Body Mass Index (BMI) between 25-35 kg/m2;
* Diagnosed T2DM (subjects are allowed to use oral antidiabetics and/or to be on a diabetes diet) or impaired glucose tolerance (defined as blood glucose > 7.8 mmol/l and < 11.0 mmol/L, two hours after ingesting 75 gram glucose in 150 ml water)

Exclusion Criteria:

* known allergy to (chicken) egg proteins;
* active cardiovascular diseases like congestive heart failure or recent (< 6 months) event (acute myocardial infarction, cerebral vascular incident);
* severe medical conditions related to the intestine that might interfere with the study such as inflammatory bowel disease and celiac disease;
* the use of insulin;
* the use of medication such as antihypertensives, statins or drugs that change gastric motility or emptying;
* abuse of drugs or alcohol (> 21 units per week);
* pregnant or breast-feeding women;
* current smoker;
* having donated blood at the blood bank within a period of 8 weeks prior to the start of the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-09; Primary Completion 2013-05 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
The change (baseline vs 2 hours, and baseline vs 2 days) in arterial stiffness measured as carotid-femoral pulse wave velocity | baseline vs 2 hours, baseline vs 2 days

SECONDARY OUTCOMES:
Changes in glucose and insulin concentrations and calculated HOMA-index, incretins, lipids, characteristics of the microcirculation, and non-invasively assessed upper-arm blood pressure and central aortic systolic blood pressure and heart rate changes | baseline vs 2 hours, and baseline vs 2 days

CONTACTS AND LOCATIONS:
Overall Officials: Jogchum Plat, Dr., Principal Investigator — Maastricht University
Locations (1):
- PreCare Trial & Recruitment, Beek, Limburg, Netherlands